CLINICAL TRIAL: NCT06071793
Title: Family Integration in Therapy Activities in the Intensive Care Unit: The FIT-ICU Feasibility Study
Acronym: FIT-ICU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Kimberley Lewis, Assistant Professor, Intensivist, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15669
Record Dates: First submitted 2023-09-19; First posted 2023-10-06 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Critical Illness; Delirium
MeSH Terms: conditions — Critical Illness; Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): Patients to receive mobility interventions from trained family members
  Interventions: Other: Family involvement

INTERVENTIONS:
Other: Family involvement — Family delivery of mobility activities

SUMMARY:
An ICU admission is stressful for not only patients but their families as well. Research has shown that involving family members during a loved one's ICU stay can be helpful for them, but there is not clear direction on the best way to do this. For patients, family presence as well as early movement during their ICU stay has been shown to help recovery from things like delirium (a state of confusion) faster, and might prevent the weakness that can happen with a stay in the ICU. In this study, the investigators will explore whether having family help with moving patients through physiotherapy guided exercise can help both patients and families have a better experience and result from their ICU stay.

The investigators hypothesize that family involvement in activities as part of an overall physiotherapy treatment plan will provide a tangible means for family members to engage in the care of their critically ill loved one, thus improving outcomes for both critically ill patients and family members.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) in the ICU
* Anticipated length of stay ≥48 hours for whom a request for physiotherapy has been placed by the treating physician
* Appropriateness for physiotherapy confirmed by the unit's physiotherapist.
* Families will be eligible if they are able to be present in ICU during physiotherapist or research team work hours until they are cleared to deliver activities independently, then at least three times weekly thereafter.

Exclusion Criteria:

* Patients who are receiving end of life care
* Patients who have high risk injuries including spinal cord injury or spinal fractures, post-operative from spinal surgery, and untreated hip or long bone fractures
* Patients at risk of raised intracranial pressure (ICP) (e.g. Malignant middle cerebral artery stroke, large subarachnoid hemorrhage), admitted post trauma activation, post-operative from brain surgery or with external ventricular drain (EVD) in situ.
* Patients who are bed-bound or require mechanical lift at baseline who would not otherwise be offered physiotherapy services.
* Exclusion criteria for families include any major barriers to participation, i.e., physical, cognitive, emotional or capacity to understand and communicate with the team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility - consent rate | Study duration - up to one year
  We define a successful consent rate as > 70% of SDMs or patients approached to consent, agreeing to take part in the study
Feasibility - recruitment rate | Study duration - up to one year
  We define a successful recruitment rate as achieving enrolment of four patients per month over the duration of the trial
Feasibility - protocol adherence | During ICU stay, censored at 1 month
  We define successful adherence as average family involvement in ≥ 3 sessions/week. Furthermore, adherence to documentation of involvement will be successful if documented by family for ≥80% of sessions
Feasibility - resources | Study duration - up to one year
  Physiotherapist and nurse outcomes will include inability to train families due to physiotherapy or team resources, and number of sessions per week cancelled due to inadequate staffing resources during the patients ICU stay.

SECONDARY OUTCOMES:
Patient Delirium | During ICU stay, censored at 1 month
  CAM-ICU
Patient & Family PTSD symptoms | 1 & 3 months
  IES-R
Adverse Events | During ICU stay, censored at 1 month
  Falls, hypotension, bradycardia, line removal, unplanned extubation, inappropriate family intervention, unexpected injuries
Family satisfaction | 1 & 3 months
  23-item Family Satisfaction in the ICU questionnaire; HADS scale

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley Lewis, MD, Principal Investigator — The Research Institute of St Joe's Hamilton; Laiya Carayannopoulos, MD, Principal Investigator — The Research Institute of St Joe's Hamilton
Locations (3):
- Canada (3):
  - Brant Community Healthcare System, Brantford, Ontario
  - St Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No